CLINICAL TRIAL: NCT06727942
Title: Toward Healthy Living: Virtual Reality-Infused Treadmill Training on Aging-Related Outcomes
Brief Title: Virtual Reality-Infused Treadmill Training on Aging-Related Outcomes
Acronym: V-TARGET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Xiangli, Associate Professor, The University of Texas at Arlington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-0678; 2021-0678 (Other: University of Texas at Arlington)
Record Dates: First submitted 2024-10-18; First posted 2024-12-11 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Adult ALL
Keywords: Virtual-Reality; Fall Risk Invention; Physical Activity; Neuromotor Rehabilitation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two groups: the intervention group and the control group. All participants will exercise on the Virtuix Omni 360-degree self-paced, non-powered treadmill-simulator in the lab for 5-weeks (2 days/week, 30 minutes/session, 10 sessions total. The treadmill-simulator is a first-of-its-kind motion platform on which an individual can walk and run at a self-paced speed in 360 degrees without risk of falling or colliding with other people. The V-TARGET intervention group will self-pace their locomotor action (walking/running) on the Omni treadmill-simulator while they wear the Pico Neo 2 head-mounted display (HMD) headset and use the Neuro Rehab VR XR Therapy system to experience daily activity exercises/games, including Retail Therapy, Explore (gait training), Lunchtime Adventure, and Nature Walk. The control group will not do any VR exercise but will only complete the pre-post and 1-month follow-up assessment upon signing up the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- V-TARGET intervention group (Experimental): All participants in the V-TARGET intervention group will exercise on the Virtuix Omni 360-degree self-paced, non-powered treadmill-simulator in the lab for 5-weeks (2 days/week, 30 minutes/session, 10 sessions total. The treadmill-simulator is a first-of-its-kind motion platform on which an individual can walk and run at a self-paced speed in 360 degrees (i.e., forwards, sideways and backwards) without risk of falling or colliding with other people.
  The V-TARGET intervention group will self-pace their locomotor action (walking/running) on the Omni treadmill-simulator while they wear the Pico Neo 2 head-mounted display (HMD) headset and use the Neuro Rehab VR XR Therapy system to experience daily activity exercises/games, including Retail Therapy, Explore (gait training), Lunchtime Adventure, and Nature Walk.
  Interventions: Device: V-TARGET intervention
- The waitlist control group (No Intervention): The control group will not do any VR exercise but will only complete the pre-post and 1-month follow-up assessment upon signing up the study.

INTERVENTIONS:
Device: V-TARGET intervention — V-TARGET intervention will be delivered through a 360 degree self-paced treadmill in a university clinical laboratory for 5-weeks (2 days/week, 30 minutes/session) with total 10 sessions. The treadmill is the first-of-kind motion platform that an individual can walk and run at self-paced speed in 360 degree (i.e., forwards, sideways and backwards) without risk of falling or colliding with other people. During the V-TARGET intervention, participants will self-pace their locomotor action (walking/running) while they wear the HTC vivo headset and experience daily exercises/games augmented by the VR Therapy System. Therapy System is a library of VR exercises/games targeted on neurological rehabilitation, balance improvement training as well as cognitive therapy suited for variety of conditions, and includes various daily living simulation activities such as Retail Shopping, Gait Training, Cafeteria Experience, and Nature Walk.
  Arms: V-TARGET intervention group

SUMMARY:
Age-associated motor and cognitive deficits increase the risk of falls, a major cause of morbidity and mortality. Emerging evidence suggests that inflammatory mediators lead to impaired functional capacity and frailty in the elderly and suggests that immune system mediated inflammation in the brain play an important role in cognitive decline. Substantial literature has also demonstrated that age-targeted physical activity training are promising strategies for promoting the motor-cognitive process across the adult lifespan. Recently, the virtual reality (VR) application has been implemented in the neuropsychological rehabilitation settings suggesting that the VR-infused daily living activities may benefit the transfer of intervention outcomes and to promote autonomy in function of daily living such as cooking or grocery shopping. However, it remains unclear the effect of the VR-based exercise intervention (motor-cognitive impact) on older adults' cognitive function and fall prevention. The literature suggests that the similarity of VR exercises with real life activities may improve generalizability by extending the transfer of gains of training to everyday living and promote some aspects of quality of life in older adults. It is also unclear to what extent these aging-associated motor- cognitive changes may be affected by VR rehab games and whether systemic- and neuro-inflammation is ameliorated by this novel intervention in older adults.

This purpose of this study is to design and implement a Virtual Reality-Infused Treadmill Training on Aging-Related Outcomes (V-TARGET) intervention, focusing on adults (aged up to 75 years old). The study will compare the effects of V-TARGET intervention (self-paced treadmill-simulator exercise with VR rehab games) against a control group on motor-cognitive function, health-related quality of life (HRQOL), circulating inflammatory markers and cerebral/peripheral blood flow through this 5-week intervention (2 times/week, 30-minutes/session, 10 sessions total).

DETAILED DESCRIPTION:
A randomized controlled trial using a repeated measure design with a 1-month follow-up assessment will be employed. The study will compare the effects of V-TARGET intervention (self-paced treadmill exercise augmented by VR rehab games) against an active-control paradigm (self-paced treadmill exercise without VR rehab games) on motor-cognitive function, health-related quality of life (HRQOL), and circulating inflammatory markers through a 5-week V-TARGET intervention (2 times/week, 30-minutes/session, total 10 sessions). Specifically,

Primary Aim 1: To examine the effects of a 5-week V-TARGET intervention on motor function (i.e., balance/mobility and rate of fall), cognitive function (i.e., working memory and executive function), and HRQOL among older adults.

It is hypothesized that after controlling for socio-demographic variables (i.e., age, gender, SES, body mass index [BMI]), and physical activity history, individuals in the V-TARGET group would exhibit more improvement in the motor and cognitive function and better HRQOL after the intervention compared to individuals in the active control group. It is hypothesized that gains made by the experimental group at post-treatment would be maintained or enhanced at the 1-month follow-up.

Secondary Aim 2: To determine whether a 5-week V-TARGET intervention alters circulating inflammatory markers in older adults. Circulating levels of interferon (IFN)-γ, CXCL10, T cell IFN-γ production and cell surface expression of CXCR3 (the receptor for CXCL10) will be measured .

It is hypothesized that V-TARGET intervention will result in downregulation of the T cell/IFN-γ/CXCL10 inflammatory cascade and that these changes represent a potential biological mechanism by which the V-TARGET intervention improves motor-cognitive function in older adults with high risk of fall. It is hypothesized that gains made by the experimental group at post-treatment would be maintained or enhanced at the 1-month follow-up.

Secondary Aim 3: To examine the effects of a 5-week V-TARGET intervention on Cerebrovascular Health among older adults.

It is hypothesized that after controlling for socio-demographic variables (i.e., age, gender, SES, body mass index [BMI]), and physical activity history, individuals in the V-TARGET group would exhibit more improvement in the Cerebrovascular Health after the intervention compared to individuals in the active control group. It is hypothesized that gains made by the experimental group at post-treatment would be maintained or enhanced at the 1-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. adults aged up to 75 years old
2. able to walk independently, without use of an assistive device
3. English speaking

Exclusion Criteria:

1. self-disclosed limited mobility in joint(s) due to arthritis or other condition that would prevent participation
2. any ongoing orthopedic injury
3. cardiac surgery or any ongoing cardiovascular issues preventing participation or physical activity.
4. motor/cognitive disorders (Alzheimer's disease, Parkinson's disease, dementia, etc.)
5. use of a wheelchair

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is open to participants of all genders, including individuals who self-identify as male, female, non-binary, genderqueer, or any other gender identity. Individuals who self-identify as transgender or cisgender are welcomes. If participants' gender identity does not fit within traditional male or female categories, participation of the study is still welcomed.
Enrollment: 60 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Motor Function | Baseline & immediately following the intervention & and again at 1-month following completion of the intervention.
  The Tinetti scale measures motor function; the total score ranges from 0- 28: a total score of less than or equal to 18 indicates high risk of falling; score range 19-23 indicates moderate risk of falling; and more than or equal to 24 indicates low risk of falling.
Motor skill | Baseline & immediately following the intervention & and again at 1-month following completion of the intervention.
  The Bruininks Motor Ability Test (BMAT) is a standardized test of gross and fine motor skills for adults and older. It assesses fine motor integration, manual dexterity, coordination, balance and mobility, and strength and flexibility. Each subtest score is converted into scaled scores based on normative data.
  The total BMAT score is derived by summing the scores from each domain, which can then be compared to age-based norms. Higher scores indicate better motor abilities, while lower scores may suggest areas that could benefit from intervention or support.
Cognitive function: Multitasking test (MTT) | Baseline & immediately following the intervention & and again at 1-month following completion of the intervention.
  Cognitive function is assessed with CANTAB (Cambridge Neuropsychological Test Automated Battery) using a handheld tablet (10 x 10-inch iPad).
  Multitasking test (MTT) is a test of the participant's ability to manage conflicting information provided by the direction of an arrow and its location on the screen and to ignore task-irrelevant information. Outcome measures include response latencies and error scores.
Cognitive function: The spatial working memory (SWM) test | Baseline & immediately following the intervention & and again at 1-month following completion of the intervention.
  Cognitive function is assessed with CANTAB (Cambridge Neuropsychological Test Automated Battery) using a handheld tablet (10 x 10-inch iPad). The spatial working memory (SWM) test requires retention and manipulation of visuospatial information, and provides a measure of strategy as well as working memory errors. Outcome measures include errors and strategies.

SECONDARY OUTCOMES:
Circulating inflammatory markers: percentage of T cells expressing CXCR3 | Baseline & immediately following the intervention & and again at 1-month following completion of the intervention.
  Following a blood draw (~5ml or 1 teaspoon), T cell CXCR3 (the receptor for CXCL10) expression will be assessed by the standard Flow cytometry and calculated in %.
Circulating inflammatory markers: interferon-gamma (IFN-γ) | Baseline & immediately following the intervention & and again at 1-month following completion of the intervention.
  Following a blood draw (~5ml or 1 teaspoon), interferon-gamma (IFN-γ) is assessed by enzyme-linked immunoassay (ELISA) and calculated in pg/ml.
Circulating inflammatory markers: Circulating CXCL10 | Baseline & immediately following the intervention & and again at 1-month following completion of the intervention.
  Following a blood draw (~5ml or 1 teaspoon), Circulating CXCL10 is assessed by enzyme-linked immunoassay (ELISA) and calculated in pg/ml
Cerebrovascular Health: Heart Rate | Baseline & immediately following the intervention & and again at 1-month following completion of the intervention.
  Heart Rate (beats per minute): Standard heart rate measurement using electrocardiogram
Cerebrovascular Health: Systolic arterial blood pressure in the brachial artery (mmHg) | Baseline & immediately following the intervention & and again at 1-month following completion of the intervention.
  Systolic arterial blood pressure in the brachial artery (mmHg): Standard blood pressure measures
Cerebrovascular Health: Diastolic arterial blood pressure in the brachial artery (mmHg) | Baseline & immediately following the intervention & and again at 1-month following completion of the intervention.
  Diastolic arterial blood pressure in the brachial artery (mmHg): Standard blood pressure measures
Cerebrovascular Health: mean arterial blood pressure in the brachial artery (mmHg) | Baseline & immediately following the intervention & and again at 1-month following completion of the intervention.
  mean arterial blood pressure in the brachial artery (mmHg): Standard blood pressure measures
Cerebrovascular Health: Endothelial Function (% change of brachial artery diameter) | Baseline & immediately following the intervention & and again at 1-month following completion of the intervention.
  Endothelial Function (% change of brachial artery diameter): Flow Mediated dilation of the brachial artery
Cerebrovascular Health: Cerebral blood velocity (centimeters / second) | Baseline & immediately following the intervention & and again at 1-month following completion of the intervention.
  Cerebral blood velocity (centimeters / second): Measures of blood velocity on the middle cerebral artery using trans-cranial Doppler ultrasound
Health-related quality of life (HRQOL) | Baseline & immediately following the intervention & and again at 1-month following completion of the intervention.
  The SF-36 Health Survey is used to measure generic health status and HRQOL. The SF-36 comprises eight health scales: physical functioning (PF; ten items), role limitations due to physical problems (RP; four items), bodily pain (BP; two items), general health (GH; five items), vitality (VT; four items), social functioning (SF; two items), role limitations due to emotional problems (RE; three items), and mental health (MH; five items). The scores range from 0 to 100, with higher scores indicating better functional health and well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangli Gu, Principal Investigator — University of Texas at Arlington
Locations (1):
- University of Texas at Arlington Movement & Physical Activity Epidemiology Laboratory, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) may not be shared due to concerns related to participant privacy and confidentiality. While efforts are made to de-identify all data, the sensitive nature of the information collected in this study could potentially lead to the identification of participants if shared publicly. Additionally, current consent forms do not explicitly allow for the sharing of individual data outside of the research team.
  If future updates to consent or data protection protocols allow for IPD sharing, and with appropriate safeguards in place, it may be reconsidered to share IPD under controlled access conditions. For now, only aggregated data and study results will be shared to maintain the privacy of our participants.

REFERENCES:
- See also: Virtual Reality Rehab-Therapy on Neuromotor Function and Cardiovascular Health — https://mpaelab.uta.edu/research/v-rate/